CLINICAL TRIAL: NCT00561028
Title: Prevalence of Chlamydia Pneumoniae and Mycoplasma Pneumoniae in Different Forms of Obstructive Coronary Artery Disease
Brief Title: Chlamydia and Mycoplasma in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Hospital de Base (Other)
Collaborators: University of Sao Paulo (Other)
Other Study IDs: 5105/2001; 885/02
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Chlamydia Infections; Mycoplasma Infections
Keywords: Atherosclerosis; Coronary artery disease; Chlamydia pneumoniae; Mycoplasma pneumoniae
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Chlamydia Infections; Mycoplasma Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample - serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: ST-elevation acute myocardial infarction.
  Interventions: Other: blood sample analysis - mycoplasma and chlamydia antibodies
- 2: high-risk unstable angina or non-ST-elevation myocardial infarction.
  Interventions: Other: blood sample analysis - mycoplasma and chlamydia antibodies
- 3: known coronary artery disease, either asymptomatic or with stable angina.
  Interventions: Other: blood sample analysis - mycoplasma and chlamydia antibodies
- 4: blood donors without known coronary artery disease.
  Interventions: Other: blood sample analysis - mycoplasma and chlamydia antibodies

INTERVENTIONS:
Other: blood sample analysis - mycoplasma and chlamydia antibodies — Anti-Chlamydia and anti-Mycoplasma IgG antibodies were measured by indirect immunofluorescence at baseline (24 hours of hospitalization) and after 6 months (follow-up).

SUMMARY:
To test the association between anti-Chlamydia serum titers and anti-Mycoplasma antibodies with Acute Coronary Syndromes.

DETAILED DESCRIPTION:
One hundred and twenty-six patients were divided into 4 groups: Acute Coronary Syndrome with ST-elevation, Non-ST-elevation, stable coronary artery disease, and individuals without coronary disease. Anti-Chlamydia and anti-Mycoplasma IgG antibodies were measured at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yrs
* Males and females
* Agreed to sign the informed consent

Exclusion Criteria:

* Refusal to sign the informed consent
* Follow-up not possible
* For the "acute" groups, time between the pain beginning and randomization >24 hours
* Active infections
* Use of antimicrobial agents within the last 30 days
* End-stage diseases with life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 and 2 - selected after admission in coronary care unit. Group 3 - selected from out-patient cardiology clinic. Group 4 - selected from the blood donation unit.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2002-03; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that patients with acute coronary syndromes have higher levels of Chlamydia pneumonia and Mycoplasma pneumonia antibodies in comparison with patients with stable coronary artery disease or controls. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Nicolau, MD, pHD, Study Director — University of Sao Paulo

REFERENCES:
- [Derived] Maia IL, Nicolau JC, Machado MN, Maia LN, Takakura IT, Rocha PR, Cordeiro JA, Ramires JA. Prevalence of Chlamydia pneumoniae and Mycoplasma pneumoniae in different forms of coronary disease. Arq Bras Cardiol. 2009 Jun;92(6):405-11, 422-8, 439-45. doi: 10.1590/s0066-782x2009000600005. English, Multiple languages. PMID 19629306